CLINICAL TRIAL: NCT04644562
Title: The Anaesthetic and Analgesic Efficacy of Ultrasound-guided Lumbar Erector Spinae Plane Block in Patients Undergoing Lower Limb Vascular Surgery
Brief Title: Ultrasound-guided Lumbar Erector Spinae Plane Block in Patients Undergoing Lower Limb Vascular Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, doaa rashwan, Assistant professor Doaa Rashwan, Beni-Suef University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: FMBSUREC/05072020/Abd El Badei
Record Dates: First submitted 2020-07-17; First posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Anesthesia, Local

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients undergoing Lower Limb vascular Surgery (Experimental): Ultrasound-guided lumbar Erector Spinae plane block in patients undergoing Lower Limb vascular Surgery
  Interventions: Other: Erector Spinae plane block

INTERVENTIONS:
Other: Erector Spinae plane block — Ultrasound-guided lumbar Erector Spinae plane block in patients undergoing Lower Limb vascular Surgery

SUMMARY:
the investigatots hypothesized that by injection a larger volume and higher concentration of local anesthetic in lumbar erector spinae plane block could result in successful anesthesia in patient undergoing lower limb vascular surgery.

ultrasound-guided lumbar erector spinae plane block in patient undergoing lower limb vascular surgery with higher concentration of local anesthetic to asses it is efficacy as a sole anesthetic technique, it is safety and efficacy in maintaining intraoperative hemodynamics, intra and postoperative pain control .

DETAILED DESCRIPTION:
The patients will placed in lateral position. After aseptic preparation of the skin and probe, a high-frequency linear ultrasound transducer will move about 3 cm laterally on the parasagittal plane to visualize the transverse process of the (L2) vertebra. An 18-guage tuohy needle will be approached in-plane lateral to medial. When the needle initially touched the transverse process of L3 vertebrae, the needle will be gently withdrawn and hydrodissection of the plane achieved, lifting the erector spinae muscle. A 20-guage catheter will be introduced through the needle and total length inserted will be 3 cm more than the tip of needle (. 25 mL of 0.5% bupivacaine ( in increments slowly after negative aspiration will be injected in the interfascial plane observing the anesthetic spread.

Sensory and motor block will be evaluated and surgery will begin only after adequate block , if failed, general anesthesia will induced by injecting 1.5-2 mg/kg propofol, 2 μg/kg fentanyl & 0.5 mg/kg atracurium.

The patients will be ventilated via face mask with 100 % oxygen at a rate of 4 L/min and isoflurane 1.2 %. After 3 minutes, the patients will be intubated using appropriate sized cuffed oral tube lubricated with lidocaine jelly 2 % .

Maintenance of anesthesia will done using isoflurane 1.2 % in 100 % O2. Muscle relaxation will be continued by atracurium 0.1 mg/kg every 20 min. All patients will be mechanically ventilated to maintain end-tidal carbon dioxide between 35-40 mmHg. For 5 minutes, no surgical interventions will be allowed in the subjects to assess target blood pressure.

ELIGIBILITY:
Inclusion Criteria:

- ASA II and III male and female patients undergoing lower limb vascular surgery

Exclusion Criteria:

* Contraindications for regional blocks (eg. Patient refusal Infection at the injection site, coagulopathy)
* allergic reaction to drugs.
* opium addiction, any drug or substance abuse and chronic treatment with opium, non-steroidal anti-inflammatory drugs

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2020-11-20 (Estimated); Primary Completion 2021-01-30 (Estimated); Study Completion 2021-01-30 (Estimated)

PRIMARY OUTCOMES:
motor block block level | baseline, pre-intervention/procedure/surgery
  motor power

CONTACTS AND LOCATIONS:
Overall Officials: doaa rashwan, md, Principal Investigator — Beni-Suef University
Locations (1):
- Benisuef univercity, Banī Suwayf, Benisuef, Egypt

IPD SHARING:
Plan to Share IPD: Undecided